CLINICAL TRIAL: NCT06108739
Title: Randomized Trial of Anti-thymocyte Globulin Plus Low-dose Post-transplant Cyclophosphamide for GVHD Prevention in Haploidentical Donor HCT
Brief Title: ATG Plus Low-dose PT-Cy for GVHD Prevention
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommended halting the study owing to futility after the first interim analysis in August 2024.
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG plus PT-Cy in haplo-SCT
Record Dates: First submitted 2023-10-22; First posted 2023-10-31 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-08

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ATG-PTCy cohort (Experimental): The conditioning regimen is ATG/G-CSF based protocol (the so-called Beijing protocol). The rabbit ATG (Sangstat-Genzyme) 2.5mg/kg/day i.v., on days from - 5 to - 2 were administered.Two doses of 14.5 mg/kg Cy were given on days 3 and 4 post-HCT in ATG-PTCy cohort.
  Interventions: Drug: Cyclophosphamid; Drug: ATG
- ATG cohort (Active Comparator): The conditioning regimen is ATG/G-CSF based protocol (the so-called Beijing protocol). The rabbit ATG (Sangstat-Genzyme) 2.5mg/kg/day i.v., on days from - 5 to - 2 were administered.
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: Cyclophosphamid — A total of 10mg/kg ATG was administered, and two doses of 14.5 mg/kg Cy were given on days 3 and 4 post-HCT in ATG-PTCy cohort.
  Arms: ATG-PTCy cohort
Drug: ATG — A total of 10mg/kg ATG was administered.

SUMMARY:
During the past decades, the wider application of easily available haploidentical donor hematopoietic cell transplant (haplo-HCT) has been made possible through the T cell-replete (TCR) regimens including T cell regulation with anti-thymocyte globulin (ATG)/granulocyte colony-stimulating factor (GCSF) and post-transplant cyclophosphamide (PTCy). To achieve decreased non-relapse mortality (NRM) and improved long-term outcomes in haploidentical transplant, the joint use of ATG and PTCy might effectively reduce graft versus host disease (GVHD) and mortality associated with severe forms of GVHD. Recently, investigators established a regimen using low-dose PTCy in conjunction with standard-dose ATG in order to lower the risk of GVHD without compromising engraftment and disease relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute leukemia and/or myelodysplastic syndrome undergoing their first allogeneic hematopoietic stem cell transplantation;
2. Male or female , aged 12-55 years;
3. Haploidentical donor transplantation;
4. ECOG score ≤3; The basic organ function tests met the following standards;

1) Cardiac ejection index >55% 2) Creatinine ≤1.5 times the highest normal value (ULN)

Exclusion Criteria:

1. Severe brain, heart, kidney or liver dysfunction;
2. Refractory malignant state;
3. Patients with other malignant tumors requiring treatment;
4. Clinically uncontrolled severe active infection;
5. The expected survival time was less than 3 months.
6. A history of severe anaphylaxis.
7. Pregnant or lactating women;
8. Any condition considered by the investigators to be unsuitable for enrollment.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of acute graft versus host disease. | 100 days post HSCT.
  The incidence of acute graft versus host disease. The severity of acute GVHD was evaluated according to standard international criteria.

SECONDARY OUTCOMES:
Engraftment | 30 days post HSCT.
  Myeloid engraftment was defined as the first of three consecutive days with an ANC X0.5≥10^9/L.
The incidence of chronic GvHD | 1 year post HSCT.
  The incidence of chronic GvHD.
The incidence of non-relapse mortality | 1 year post HSCT.
  The incidence of non-relapse mortality
The incidence of infection | 1 year post HSCT.
  The incidence of infection
The incidence of relapse | 1 year post HSCT.
  The incidence of relapse
Overall survival | 1 year post HSCT.
  Overall survival
Disease free survival | 1 year post HSCT.
  Disease free survival
GvHD relapse free survival | 1 year post HSCT.
  GvHD relapse free survival
Immune reconstitution | 1 year post HSCT.
  Immune reconstitution was evaluated at 1, 2, 3, 6, 9 and 12 months by analysis of peripheral blood MNCs detecting CD3, CD4, CD19 and immunoglobulin (Ig) A, G and M levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Derived] Xu ZL, Han TT, Zhu XL, Liu J, Lv M, Sun YQ, Mo XD, Cheng YF, Xu LP, Zhang XH, Huang XJ, Wang Y. Randomized trial of anti-thymocyte globulin plus lowdose post-transplant cyclophosphamide to prevent graft-versus- host disease in haploidentical transplantation. Haematologica. 2025 Dec 1;110(12):2965-2973. doi: 10.3324/haematol.2025.287504. Epub 2025 Jun 19. PMID 40534493